CLINICAL TRIAL: NCT06933784
Title: Expression of Wnt5a and WNT Coreceptor (LRP5) Levels in Stage III Periodontitis Patients
Brief Title: Evaluation of Wnt5a and LRP5 Levels in Serum and Saliva Samples and the Relationship Between Clinical Periodontal Parameters
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Zulal Deniz Guner, Sub-Investigator, Ankara University
Other Study IDs: 36290600/02/2024; 1919B012324587 (Other Grant/Funding Number: The Scientific and Technological Research Council of Türkiye (TÜBİTAK))
Record Dates: First submitted 2025-04-09; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Periodontal Disease; Periodontitis (Stage 3); Periodontitis Stage III
Keywords: Wnt5a; LRP5; periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stage III periodontitis Grade B: Individuals exhibiting pocket depths of >3 mm in at least two non-adjacent teeth, radiographic evidence of alveolar bone loss extending to the middle or apical third of the root, and tooth loss of ≤4 due to periodontitis were classified as having Stage III periodontitis. The additional criterion for Grade B classification was defined as a % bone loss/age ratio of 0.25-1.
- Periodontally healthy: Individuals with no signs of alveolar bone loss and an overall oral bleeding score <10% were categorized as periodontally healthy.

SUMMARY:
Objectives: Wnt5a is a secreted Wnt ligand that plays an important role in cellular homeostasis. Wnt interaction with coreceptor low-density lipoprotein receptor-related protein 5 (LRP5) induces the proliferation of osteoblasts and prolongs their functional life. The aim of this study is evaluating the levels of Wnt5a and LRP5 in serum and saliva samples and relationship between clinical periodontal parameters.

Method: Saliva and serum samples were collected from 20 systemically healthy patients with stage III periodontitis and 20 periodontally healthy controls. Wnt5a and LRP5 levels were measured using enzyme-linked immunosorbent assay (ELISA). Clinical periodontal parameters including plaque index (PI), probing pocket depth (PPD), bleeding on probing (BOP), and clinical attachment level (CAL) were recorded.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old,
* At least 16 permanent teeth except 3rd molars,
* Individuals who do not use orthodontic appliances,
* Individuals who are not pregnant or lactating,
* Individuals without any systemic disease that may affect periodontal health,
* Systemically healthy individuals,
* Individuals who have not used anti-inflammatory and/or anti-microbial drugs in the last 6 months,
* Individuals who have not received periodontal treatment in the last 1 year

Exclusion Criteria:

* Pregnant/lactating individuals,
* Individuals who have used anti-inflammatory and/or anti-microbial drugs in the last 6 months,
* Individuals who have undergone periodontal treatment in the last 1 year,
* Individuals with psychiatric illness,
* Individuals with any oral infection,
* Individuals with <16 teeth, excluding molars,
* Individuals with alcohol dependence,
* Individuals with active infectious disease (acute hepatitis, AIDS, tuberculosis), cancer or any systemic condition that may affect periodontal tissues,
* Individuals receiving treatment with drugs known to affect periodontal tissues (phenytoin, cyclosporine A, calcium channel blockers)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients with stage III periodontitis and periodontally healthy patients admitted to Ankara University Faculty of Dentistry Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Wnt5a | 1 month
  Wnt5a is synthesized by activated antigen-presenting cells and its expression is induced by mycobacterial cell wall components and endotoxin in human antigen-presenting cells, and Wnt5a signaling is required for the overall inflammatory response of human macrophages during sepsis.The levels of Wnt5a in both serum and saliva samples were determined using commercially available ELISA kits. All assays were conducted according to the manufacturers' instructions.
LRP5 | 1 month
  Low-density lipoprotein (LDL) receptor-related protein 5 (LRP5) is a WNT coreceptor in the LRP superfamily involved in a wide range of biological processes including endocytosis, cellular communication, lipid homeostasis and embryonic development. The levels of LRP5 in both serum and saliva samples were determined using commercially available ELISA kits. All assays were conducted according to the manufacturers' instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Faculty of Dentistry, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guney Z, Kurgan S, Onder C, Tayman MA, Gunhan O, Kantarci A, Serdar MA, Gunhan M. Wnt signaling in periodontitis. Clin Oral Investig. 2023 Nov;27(11):6801-6812. doi: 10.1007/s00784-023-05294-7. Epub 2023 Oct 10. PMID 37814163
- [Background] Zhao Y, Zhang C, Huang Y, Yu Y, Li R, Li M, Liu N, Liu P, Qiao J. Up-regulated expression of WNT5a increases inflammation and oxidative stress via PI3K/AKT/NF-kappaB signaling in the granulosa cells of PCOS patients. J Clin Endocrinol Metab. 2015 Jan;100(1):201-11. doi: 10.1210/jc.2014-2419. PMID 25303486
- [Background] Williams BO, Insogna KL. Where Wnts went: the exploding field of Lrp5 and Lrp6 signaling in bone. J Bone Miner Res. 2009 Feb;24(2):171-8. doi: 10.1359/jbmr.081235. PMID 19072724